CLINICAL TRIAL: NCT06494124
Title: Comparison of Efficacy and Safety of Transcranial Alternating Current Stimulation vs Transcranial Direct Current Stimulation on Psychopathology Measures and Neurocognition in Chronic Schizophrenia: A Randomized Double-blind Controlled Trial
Brief Title: Efficacy and Safety of tACS vs tDCS in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, BISWA RANJAN MISHRA, Additional Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T/EMF/Psych/21/67
Record Dates: First submitted 2024-04-03; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The intervention arms are Experimental (tACS), Active comparator (tDCS) and control comparator (sham). The patients in all 3 arms will continue to receive the ongoing antipsychotics.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tACS group (Experimental): 10 Hz 2 mA peak-to-peak stimulation will be for 20 minutes, at zero-degree phase difference and zero offset current
  Interventions: Device: transcranial Alternating current stimulation (tACS)
- tDCS group (Active Comparator): tDCS stimulation: 2 mA stimulation will be applied for 20 minutes
  Interventions: Device: transcranial Direct current stimulation (tDCS)
- sham controlled group (Sham Comparator): 1mA current will be applied for the first 30 seconds, to provide the initial sensation of real stimulation and then the current will be stopped, thus minimizing the stimulatory effects
  Interventions: Device: Sham controlled

INTERVENTIONS:
Device: transcranial Alternating current stimulation (tACS) — It is a non-invasive brain stimulation technique that uses small, pulsed alternating current (1mA) to modulate lasting cortical excitability, producing facilitatory or inhibitory effects upon a variety of behaviours, with proven efficacy in various neuropsychiatric disorders.
  Arms: tACS group
Device: transcranial Direct current stimulation (tDCS) — It is a non-invasive brain stimulation technique that uses constant, low direct current to modulate lasting cortical excitability, producing facilitatory or inhibitory effects upon a variety of behaviours, with proven efficacy in various neuropsychiatric disorders.
  Arms: tDCS group
Device: Sham controlled — 1mA current will be applied for the first 30 seconds to provide the initial sensation of real stimulation, and then the current will be stopped, thus minimizing the stimulatory effects. It is known to have no effect on psychopathology/neuro-cognition and means to mimic the tDCS/tACS (in order to help blinding of the participants).
  Arms: sham controlled group

SUMMARY:
This clinical trial aims to compare the efficacy and safety of transcranial Alternating current stimulation (tACS) vs. transcranial Direct current stimulation (tDCS) vs. sham stimulation in chronic schizophrenia.

The main question it aims to answer is:

• In comparison to tDCS, can tACS improve the clinical outcome of patients with chronic schizophrenia?

Participants will be randomised into 3 groups receiving either tDCS, tACS or sham stimulation and changes in psychopathology and neuro-cognition with the interventions will be compared within and between the groups. The primary outcome measure is the Positive and Negative Syndrome Scale (PANSS), while secondary outcome measures are the Auditory Hallucination Rating Scale (AHRS), Brief Cognitive Assessment Tool for Schizophrenia (B-CATS), and Global Assessment of Functioning (GAF).

DETAILED DESCRIPTION:
The proposed double-blind RCT will be conducted over 3 years involving 2 centres among patients with chronic schizophrenia (moderate-severe symptoms) of either gender, aged between 18 and 60. Those with any psychiatric emergency or contraindications for tDCS will be excluded. At baseline, PANSS will be administered to assess the severity of symptom dimension, AHRS for auditory hallucinations, B-CATS for neurocognitive deficits and GAF for global functionality. Patients will be randomized equally to 3 treatment groups: tACS, tDCS, or sham stimulation (30 in each group). The intervention will involve Cathodal stimulation of left TPJ and Anodal stimulation of left DLPFC. The transcranial brain stimulations: tACS, tDCS, or sham stimulation, will be given 2 sessions per day for 10 days. Following the 5th day and after the last treatment session, PANSS, AHRS, B-CATS, and GAF will be readministered to observe for the changes in the various outcome parameters. Any new treatment-emergent serious adverse effect will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Schizophrenia as per ICD-10 DCR for more than 2 years
2. Moderate-severe symptoms (PANSS score > 75 and/or CGI-SCH score>4) [24]
3. On stable dosing of antipsychotic medications (no changes in medication or doses for 1 month prior to enrolment)
4. Both sexes; Age range: 18-60 years
5. Right-handed
6. Written informed consent by the patient

Exclusion Criteria:

1. Features suggestive of psychiatric emergency (for example: suicidal risk, catatonia, prolonged nutritional deprivation) or others (for example: aggression or excitement)
2. Any contraindication to tDCS procedure: Metal in the head, Implanted brain medical devices, Local lesion or injury in the scalp / head
3. Co-morbid neurological disease
4. Left Handed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Baseline, Day 5, Day 10
  Measures psychopathology and illness severity in schizophrenia

SECONDARY OUTCOMES:
Auditory Hallucination Rating Scale (AHRS) | Baseline, Day 5, Day 10
  Measures severity of auditory hallucinations in schizophrenia
Brief Cognitive Assessment Tool for Schizophrenia (B-CATS) | Baseline, Day 5, Day 10
  Measures neurocognitive deficits in schizophrenia
Global Assessment of Functioning (GAF) | Baseline, Day 5, Day 10
  Measures overall functioning of the patients with mental illness including schizophrenia

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Scinces - Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No